CLINICAL TRIAL: NCT03914261
Title: Expanded Access to Risankizumab
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C19-882
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Crohn's Disease; Ulcerative Colitis (UC)
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — risankizumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Risankizumab — Tablet
  Other Names: ABBV-066; BI 655066

SUMMARY:
This is an expanded access program (EAP) for eligible participants with Crohn's Disease (CD). This program is designed to provide access to risankizumab, prior to approval by the local regulatory agency, to patients with the highest unmet need and an urgent need for treatment, where risankizumab may prolong survival, prevent occurrence of clinical events associated with significant morbidity and/or mortality, or stabilize a progressive debilitating disease. Availability will depend on a review of the eligibility of the patient and local approval status of risankizumab for CD. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie